CLINICAL TRIAL: NCT06960187
Title: Piloting Resilience Focused Mental Health Intervention (Weyera) With Ethiopian and Eritrean Youth
Brief Title: Weyera Mental Health Pilot Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Sophia Hussen, Associate Professor of Public Health and Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008231; R21MD019304-01A1 (NIH)
Record Dates: First submitted 2025-04-08; First posted 2025-05-07 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Mental Health Issue
Keywords: Eritrean origin; Ethiopian; Psychoeducation; Coping skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Other): Participants enrolled in the intervention group will begin the intervention 1-2 weeks after group assignment and will complete a baseline survey before the start of the intervention, satisfaction surveys at the end of each session, and an endline survey. At the end of the intervention, a subset of participants will also take part in in-depth interviews
  Interventions: Behavioral: Weyera Intervention
- Wait-List Control Group (Other): A wait-list control design ensures the ethical treatment of participants by guaranteeing that all individuals will have access to the potentially impactful intervention after a brief waiting period. Participants in the wait-list control group will begin the full intervention starting at month 4 following their enrollment.
  Interventions: Behavioral: Delayed intervention (waitlist control)

INTERVENTIONS:
Behavioral: Weyera Intervention — Weyera intervention is an eight-week program featuring weekly, two-hour facilitated group sessions with 6-10 participants in each group, led by trained lay facilitators. Each session will address the weekly topic and introduce an evidence-based coping strategy (e.g., mindfulness, positive refocusing) that participants can practice over the following week. Within this outline, we will create intervention activities based on theory-based change methods and practical applications matched to objectives and determinants in the Logic Model of Change.
  Outline of major modules for the eight weeks:
  1. Introduction to mental health
  2. Stress and family pressure
  3. Self-exploration and critical reflection
  4. Intersectional Identities
  5. Family Relationships
  6. Discussing mental health in the Ethiopian and Eritrean communities
  7. Trauma and Abuse
  8. Navigating mental health services
  Arms: Intervention
Behavioral: Delayed intervention (waitlist control) — Wait-list control participants will be assigned to a group for initiation of the full intervention beginning at month 4 after their enrollment (i.e., beginning after they, and their corresponding intervention group, have completed their intervention and two follow-up surveys). Wait-list control participants will complete surveys at enrollment (baseline), 2 months (pre-intervention), 4 months (pre-intervention), 6 months (immediate post-intervention), and 8 months (post-intervention).
  Arms: Wait-List Control Group

SUMMARY:
This study aims to pilot a group-level intervention focused on mental health and resilience among Ethiopian and Eritrean youth. The study follows previous work that showed high rates of mental health outcomes (depression, anxiety, post-traumatic stress disorder (PTSD)) among Ethiopian and Eritrean youth in Atlanta. The goal is to determine the acceptability, feasibility, and safety of this culturally relevant group-level intervention before a larger trial to improve resilience processes that support mental wellness in a community-based setting.

DETAILED DESCRIPTION:
The goal of this study is to develop and pilot test a Wellness: Ethiopian/Eritrean Youth Exploring Resilience and Awareness (Weyera), mental health-focused, culturally targeted, group-level intervention. This intervention aims to provide psychoeducation, develop coping skills, and create a space for open discussion.

The study will use a waitlist control design, recruiting participants randomly assigned to either the intervention or control (delayed intervention) group.

Participants will attend 8 weekly sessions (~2 hours each) that include psychoeducation, interactive activities, and coping skills practice. Sessions will be facilitated by trained community health workers. Participants will also complete baseline and follow-up surveys at 2-, 4-, and 6-month post-enrollment, as well as post-session evaluation surveys after each session.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 29 years old
* Ethiopian and/or Eritrean ethnicity by self-report
* Able to read and understand English
* Resident of Atlanta Metropolitan Statistical Area
* Available and interested to participate in 2-hour weekly sessions over 8 weeks and complete relevant surveys

Exclusion Criteria:

* Age < 18 or > 29 years old
* Unwilling or unable to provide informed consent.
* Not a resident of the Atlanta Metropolitan Statistical Area

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Satisfaction Survey | 2 months (immediate post-intervention survey), 4 months (post-intervention), 6 months (endline).
  Acceptability will be measured using satisfaction surveys at the end of each session.
Acceptability of the intervention is a subset of participants | 6 months (endline).
  A subset of participants will complete qualitative interviews: Open-ended questions at the end of the study. There is no measuring scale for these interviews.
Recruitment Rates | 2 months (immediate post-intervention survey), 4 months (post-intervention), 6 months (endline).
  Feasibility will be measured by monitoring the recruitment rate (the number of screenings conducted, along with the proportion of eligible individuals who agree to enroll).
Retention | Baseline, 2 months (immediate post-intervention survey), 4 months (post-intervention), 6 months (endline).
  Retention of participants throughout the 8 sessions will be monitored using attendance logs during each visit. This will help determine feasibility of the program.
Fidelity | Baseline, 2 months (immediate post-intervention survey), 4 months (post-intervention), 6 months (endline).
  Fidelity will be measured using the intervention logs to assess the extent to which the intervention components (number of sessions completed, length of sessions, topics discussed) adhere to the intervention protocol.
Adverse Events | Throughout study participation up to 6 month (endline)
  Adverse event tracking forms will be used to track any safety related issues with the intervention.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression (CES-D) Scale | Baseline, 2 months (immediate post-intervention survey), 4 months (post-intervention), 6 months (endline).
  Depression will be assessed using the CES-D scale, with the total score being the sum of the 20 questions. The possible score range is 0 to 60, with a score of 16 or higher indicating depression. Higher scores reflect a greater severity of symptoms.
Generalized Anxiety Disorder 7-item scale | Baseline, 2 months (immediate post-intervention survey), 4 months (post-intervention), 6 months (endline).
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a widely used, self-administered diagnostic tool designed to screen for and assess the severity of generalized anxiety disorder (GAD). The GAD-7 consists of seven items that measure the severity of various symptoms of GAD, with response categories assigned specific point values. The response options range from "not at all" (0 points), "several days" (1 point), "more than half the days" (2 points), to "nearly every day" (3 points), with a total score range of 0 to 21 points. Scores of 5, 10, and 15 are used as cut-off points for mild, moderate, and severe anxiety, respectively.
Posttraumatic Stress Disorder (PTSD) Checklist (PCL-5) | Baseline, 2 months (immediate post-intervention survey), 4 months (post-intervention), 6 months (endline).
  The Post-Traumatic Stress Disorder (PTSD) Checklist, commonly referred to as the PCL-5, is a widely used screening tool for diagnosing PTSD. The PCL-5 is a self-report assessment consisting of 20 items, rated on a 5-point Likert scale (0 = "Not at all" to 4 = "Extremely"). A total symptom severity score, ranging from 0 to 80, is obtained by summing the scores for each of the 20 items. Higher scores reflect a greater severity of symptoms.
Perceived social support | Baseline, 2 months (immediate post-intervention survey), 4 months (post-intervention), 6 months (endline)
  Perceived social support will be assessed using the Multidimensional Scale of Social Support, a 12-item scale that measures various aspects of social support. Each item has response categories of 1-7, with higher scores indicating higher levels of social support. A mean scale score is calculated by averaging the score for each item and categorized as follows: Low social support (1- 2.9), moderate support (3 - 5), and high support (5.1 - 7).
Affirming ethnic identity beliefs | 6 months (endline).
  This outcome will be explored using qualitative interviews upon completion of the study. There are no units of measurement
Mental Health Service Utilization assessed using a structured self-report questionnaire | Throughout study participation up to 6 month (endline)
  Mental health care-seeking attitudes, intentions, and the frequency and type of mental health services utilized by participants will be assessed using a structured, self-report questionnaire developed for this study. This is a descriptive measure and does not use a scored scale.
Perceived resilience | Baseline, 2 months (immediate post-intervention survey), 4 months (post-intervention), 6 months (endline)
  This outcome will be measured using the brief resilience scale, a 6-item scale with each item responses ranging 1 - 5. Scores are averaged across items and categorized as low resilience (1 - 2.99), normal resilience (3 - 4.3) and high resilience (4.31 - 5).

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Hussen, MD, MPH, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Rollins School of Public Health, Atlanta, Georgia
  - Ethiopian Community Association In Atlanta, Clarkston, Georgia
  - Eritrean-American Community Association of Georgia, Stone Mountain, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The research team will share the results of surveys and clinical abstracted data in a de-identified dataset.
Supporting Information: Study Protocol
Time Frame: The de-identified dataset will be available after the study and data analysis are complete.
Access Criteria: All requests accompanied by a methodologically sound proposal must be emailed to the principal investigator.